CLINICAL TRIAL: NCT07164261
Title: Effectiveness of Progressive Muscle Relaxation Training in Disaster Victims With Post-traumatic Stress Disorder: a Randomized Controlled Study
Brief Title: Progressive Muscle Relaxation Training in Post-traumatic Stress Disorder in Disasters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Mesut Arslan, assistant professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tssb-kgee
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder; progressive muscle relaxation training
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: The individuals will be divided into two groups: PGDI and Control groups using block randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PKGE GROUP (Experimental): Progressive muscle relaxation training will be given additionally to individuals in the PKGE group.
  Interventions: Other: progressive muscle relaxation training
- CONTROL GROUP (No Intervention): Individuals in the control group will continue their standard treatment.

INTERVENTIONS:
Other: progressive muscle relaxation training — Progressive muscle relaxation training will be performed twice a week, each session lasting 20-30 minutes, for a total of 12 sessions over 6 weeks.
  Arms: PKGE GROUP

SUMMARY:
This study aims to investigate the effectiveness of progressive muscle relaxation training in disaster victims experiencing post-traumatic stress disorder.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is an often devastating psychiatric condition that can occur in people who experience or witness a traumatic event.The estimated lifetime prevalence of PTSD is reported to be 6.8%.While trauma-focused psychotherapy is generally the first-line treatment in PTSD management, pharmacological treatments (selective serotonin reuptake inhibitors) are recommended in second-line treatment.Additionally, various physiotherapy and rehabilitation approaches such as aerobic, respiratory, relaxation, stretching, balance and strengthening exercises can also be used.Progressive muscle relaxation training increases parasympathetic nervous system activity. This is said to reduce anxiety and stress levels and improve sleep quality, resulting in physical and mental relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals affected by disasters
* Those diagnosed with PTSD according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria
* Aged 18-65 will be included

Exclusion Criteria:

* Individuals with uncontrolled comorbidities accompanying PTSD (such as diabetes or hypertension)
* serious psychological disorders (such as dementia, psychosis/manic episodes)
* musculoskeletal conditions that would interfere with exercise training
* received PKGE training within the last year
* pregnant
* have substance abuse
* have communication difficulties, and are unable to use technology for telerehabilitation will not be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist (PCL-5) questionnaire | Change from baseline at 6 weeks
  This is a 20-question questionnaire, valid and reliable in Turkish, that assesses PTSD symptoms as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Questions are scored from 0 to 4, and the total score ranges from 0 to 80. A score of 47 or higher indicates the presence of PTSD.
Depression Anxiety and Stress Scale-21 (DASS-21) | Change from baseline at 6 weeks
  It assesses an individual's condition over the past week. It is a 21-question survey consisting of three subscales: depression, anxiety, and stress. A high score on the scale indicates the presence and severity of depression, anxiety, and stress.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at 6 weeks
  It is a 19-item index, valid and reliable in Turkish, that assesses individuals' sleep quality and disturbances over the past month. The index's 18 scored questions consist of seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleeping pill use, and daytime dysfunction. Each component is scored on a 0-3 scale, with a total score ranging from 0 to 21. A total PSQI score greater than 5 indicates inadequate sleep quality, while scores of 6-10 indicate poor sleep, and scores of 11 or higher indicate long-term sleep disturbance.
Fatigue Severity Scale (FSS) | Change from baseline at 6 weeks
  It is a nine-item scale, valid and reliable in Turkish, that assesses individuals' fatigue levels. Individuals score each item on a scale of 1 to 7 (1 = completely disagree, 7 = completely agree). The total scale score ranges from 0 to 63, with scores of 36 and above indicating severe fatigue.
Short Form-36 (SF-36) questionnaire | Change from baseline at 6 weeks
  It is a valid and reliable questionnaire in Turkish that assesses individuals' quality of life. It consists of 36 questions and eight subscales: physical function, physical role, emotional role, pain, vitality, general health, and mental health. The total score ranges from 0 to 100, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren Universty, Bitlis, Bitlis /merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No